CLINICAL TRIAL: NCT04845724
Title: The Effect of Dietary Phosphorus Load and Food Matrix on Postprandial Serum Phosphate in Hemodialysis Patients
Brief Title: Dietary Phosphorus Load and Postprandial Serum Phosphate in HD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Joseph Eustace, Professor Joseph Eustace, University College Cork
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16-CRFC-32
Record Dates: First submitted 2021-04-11; First posted 2021-04-15 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Hemodialysis
Keywords: Dietary phosphorus; Hyperphosphatemia; Hyperkalaemia; Phytate; Hemodialysis
MeSH Terms: conditions — Hyperphosphatemia; Hyperkalemia

STUDY DESIGN:
Masking Description: Catering staff, who were blinded to the identity of the participants, provided meals in random order. Participants were blinded to the initial meal selection until the day of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Diet (Active Comparator): The standard diet was based on the current dialysis diet sheet. The standard diet main meal contained a higher proportion of foods with a higher phosphorus to protein ratio (salmon and dairy), and foods with higher phosphorus bioavailability (cake). The diet was tailored for each participant to provide 1.1g protein/kg ideal body weight. The major differences between the diets were at the main meal.
  Interventions: Other: Standard Diet
- Modified Diet (Experimental): The modified diet, representative of the proposed modified phosphorus diet used food of lower phosphorus to protein ratio such as beef and less dairy. Approximately 30% dietary phosphorus in the modified diet came from foods with significant phytate content such as pulses, nuts and whole grains. The modified diet was tailored for each participant to provide 1.1g protein/kg ideal body weight.
  Interventions: Other: Modified Diet

INTERVENTIONS:
Other: Standard Diet
  Other Names: Modified Diet
  Arms: Standard Diet
Other: Modified Diet
  Arms: Modified Diet

SUMMARY:
This study is to investigate the acute postprandial effect of a modified versus standard low phosphorus diet on serum phosphate, potassium and intact parathyroid levels in prevalent hemodialysis (HD) patients

DETAILED DESCRIPTION:
Background: Potential dietary strategies for controlling hyperphosphataemia include the use of protein sources with lower phosphorus bioavailability such as pulses and nuts, focus on phosphorus to protein ratios and the avoidance of all phosphate additives.

Method: Controlled crossover feeding study in 8 HD patients. On one day, participants were directly observed eating a standard low phosphorous diet and on the other day, a modified low phosphorus diet. The modified diet included beef and less dairy, with a lower phosphorus to protein ratio, as well as plant-based protein, whole grains, pulses and nuts containing phytates which reduces phosphorus bioavailability. Both diets were tailored for each participant to provide 1.1g protein/kg ideal body weight. Participants provided fasting bloods before breakfast, a pre-prandial sample before lunch and samples at one hour intervals for the four hours after the meal, for analysis of phosphate, potassium and intact parathyroid hormone (iPTH).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age;
* on dialysis for > 3 months;
* pre-dialysis serum phosphate < 2.5 mmol/L and
* serum potassium < 6.3 mmol/L on most recent routine monthly blood test;
* urinary outputs of < 200 ml/day by self-report;
* being in their usual state of health

Exclusion Criteria:

* history of diabetes mellitus
* history of parathyroidectomy
* history of calciphylaxis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11-26 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
Serum Phosphate | Post -prandial period (4 hours)
  mmol/l

SECONDARY OUTCOMES:
Serum Potassium | Post -prandial period (4 hours)
  mmol/l

OTHER OUTCOMES:
Serum intact Parathyroid Hormone | Post -prandial period (4 hours)
  ng/L

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Eustace, MB, Principal Investigator — University College Cork

IPD SHARING:
Plan to Share IPD: No
We did not get consent for publication of identifiable data, and so as perHrynaszkiewicz et al 2010 anthropometric data, sex, ethnicity and age will not be reported in the raw data. We will report the biochemical data and nutrient intake data which allow the reproduction of the analysis we will present.

REFERENCES:
- [Derived] Byrne F, Gillman B, Palmer B, Kiely M, Eustace J, Kearney P, Davidson F, Shiely F. The effect of dietary phosphorus load and food matrix on postprandial serum phosphate in hemodialysis patients: a pilot study. HRB Open Res. 2021 Nov 10;4:119. doi: 10.12688/hrbopenres.13382.1. eCollection 2021. PMID 35187396